CLINICAL TRIAL: NCT07305038
Title: Analysis of the Clinical Effect of EDLS-clips in Endoscopic Full-thickness Resection
Brief Title: EDLS-clips in Endoscopic Full-thickness Resection
Status: Completed | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Mingliang Feng, Associate professor, First Hospital of China Medical University
Other Study IDs: End-D-F1
Record Dates: First submitted 2025-09-24; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Gastric Submucosal Tumors; Endoscopic Full Thickness Resection (EFTR)
Keywords: endoscopic submucosal dissection; endoscopic full-thickness resection; endoscopic double-layer suturing method with metallic clips; submucosal tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: endoscopic double-layer suturing method with metallic clips — This study comprises case series of 43 patients with gastric SMTs who underwent EDLS-clips after EFTR in our center.

SUMMARY:
A retrospective analysis was conducted on patients who visited from March 2022 to May 2024 and underwent endoscopic full-thickness resection and double-layer suture with titanium clips under endoscopy. The basic clinical information, tumor characteristics, overall resection rate and postoperative complications of all patients were evaluated. To analyze the clinical effect of double-layer suture technique with titanium clips under endoscopy in clamping the wound surface after full-thickness endoscopic resection.

DETAILED DESCRIPTION:
The clinical data of patients who underwent endoscopic double-layer suture with titanium clip after endoscopic full-thickness resection at the Endoscopy Center of the First Affiliated Hospital of China Medical University from March 2022 to May 2024 were collected. Indications for endoscopic treatment of SMT: ① For tumors suspected of having malignant potential through preoperative examination or confirmed by biopsy pathology, especially for those suspected of having GIST with a preoperative long diameter of ≤2cm, low risk of recurrence and metastasis, and possibly complete resection, endoscopic resection can be performed. For suspected low-risk GIST with a tumor long diameter greater than 2cm and preoperative assessment excluding lymph node or distant metastasis, under the premise of ensuring complete tumor resection, endoscopic resection can be considered to be carried out by experienced endoscopists in units with mature endoscopic treatment techniques. ② SMT with symptoms (such as bleeding, obstruction). ③ Patients who are suspected of being benign by preoperative examination or confirmed by pathology, but cannot be followed up regularly or whose tumors increase in a short period of time during the follow-up period, or who have a strong willingness for endoscopic treatment. When the tumor protrudes into the serosa or partially grows outside the cavity, or when it is found during the operation that the tumor is closely adhered to the serosa layer and cannot be separated, EFTR can be selected for endoscopic treatment. Complications related to SMT in endoscopic treatment: (1) Intraoperative bleeding: Bleeding that causes the patient's hemoglobin to drop by more than 20g/L. (2) Postoperative bleeding: Postoperative bleeding is manifested as hematemesis, melena or hematochezia, etc. In severe cases, there may be manifestations of hemorrhagic shock. It mostly occurs within one week after the operation, but it can also appear 2 to 4 weeks after the operation. (3) Delayed perforation: It is usually manifested as abdominal distension, aggravated abdominal pain, signs of peritonitis, fever, and imaging examination shows gas accumulation or an increase in gas accumulation compared to before. (4) Gas-related complications: including subcutaneous emphysema, mediastinal emphysema, pneumothorax and pneumoperitoneum, etc. (5) Digestive tract fistula: Digestive juices caused by endoscopic surgery flow into the thoracic or abdominal cavity through the leakage channel. From a patient's medical records collected in the patient's age, gender, lesion characteristics, endoscopic treatment and postoperative clinical course details and other information. The investigators define the position of the lesion on the short axis as the position of the lesion center. The closure time is defined as the period from the start (when the investigators insert the clamp into the visual field channel) to the end of closure (when the last clamp is released).

ELIGIBILITY:
Inclusion Criteria:

1. Having a tumor located in the stomach and confirmed to originate from the muscularis propria on endoscopic ultrasonography (EUS);
2. Having a tumor diameter >1 cm, which can be completely resected using endoscopic techniques, and with low risk of residue and recurrence;
3. Preoperative assessment excluded those with lymph node or distant metastasis;
4. Being able to tolerate tracheal intubation anesthesia, with no coagulation dysfunction or anticoagulant drugs stopped before EFTR.

Exclusion Criteria:

1. Patients who have been evaluated preoperatively and are considered to have lymph node or distant metastasis;
2. who cannot tolerate general anesthesia with endotracheal intubation,
3. who have not discontinued anticoagulant drugs before EFTR or have coagulation dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study comprises case series of 43 patients with gastric SMTs who underwent EDLS-clips after EFTR in our center from March 2022 to May 2024.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
The complete closure rate of EDLS-clips | Perioperative/Periprocedural
  Successful closure refers to the full coverage of the mucosal defect by surrounding normal mucosa without any gaps.

SECONDARY OUTCOMES:
Operative time | Perioperative/Periprocedural
  Operative time refers to the duration of the entire tumor resection and suture process (from the first incision of the mucosa with the knife to the completion of wound closure).
Suturing time | Perioperative/Periprocedural
  Suturing time was defined as the period from when the operator inserts the first metallic clip through the instrument channel to close the wound until the release of the final metallic clip (for cases involving simultaneous cutting and suturing, the suturing time includes part of the tumor resection time).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Investigators share the technical operation of this endoscopic double-layer suture method for closing the wounds after endoscopic full-thickness resection (EFTR) for gastric submucosal tumors (SMTs) using endoscopic double-layer suturing method using metal clips (EDLS-clips). This study included 43 patients with gastric SMTs who received EFTR and were treated with EDLS-clips from March 2022 to May 2024 at our center. The primary outcome was the complete closure rate by EDLS-clips. Secondary outcomes included closure time, the number of clips used, and adverse events.